CLINICAL TRIAL: NCT00771407
Title: A Prospective, Multicenter, Randomized, Controlled, Third-party Blinded Study of Strattice Fascial Inlay for Parastomal Reinforcement in Patients Undergoing Surgery for Permanent Abdominal Wall Ostomies
Brief Title: Parastomal Reinforcement With Strattice
Acronym: PriSm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: LFC2008.01.01
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Parastomal Hernia
Keywords: Ostomy creation; Parastomal hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strattice fascial inlay (Active Comparator): Strattice will be placed as a fascial inlay to support the ostomy site
  Interventions: Device: Strattice Reconstructive Matrix
- Standard ostomy construction (Other): Ostomy will be created in the standard fashion
  Interventions: Other: Standard ostomy creation

INTERVENTIONS:
Device: Strattice Reconstructive Matrix — Strattice will be placed as a fascial inlay to support stoma sites
  Arms: Strattice fascial inlay
Other: Standard ostomy creation — Ostomy will be created as routinely performed
  Arms: Standard ostomy construction

SUMMARY:
The purpose of this study is to compare the clinical outcomes of patients undergoing surgery for a permanent abdominal wall ostomy with and without placement of Strattice fascial inlay, as measured by postoperative occurence of parastomal hernia.

ELIGIBILITY:
Inclusion Criteria:

* adults
* need for permanent ileostomy or colostomy

Exclusion Criteria:

* history of hernia at new ostomy site
* has previously implanted surgical mesh at site of planned ostomy
* requires a temporary ostomy
* has need for multiple ostomies
* is receiving chronic immunosuppression therapy, has MELD score of > 17, has severe COPD, systemic infection, or known collagen disorder
* is bedridden or otherwise non-ambulatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Fleshman, MD, Principal Investigator — Washington University, St Louis MO
Locations (23):
- United States (23):
  - University of South Alabama, Mobile, Alabama
  - Office of Dr Phillip Fleshner, Los Angeles, California
  - University of California at Irvine, Orange, California
  - Stanford University Medical Center, Stanford, California
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Illinois, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Louisiana State University, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - University of Maryland/Baltimore VA, Baltimore, Maryland
  - Spectrum Health - Butterworth Hospital, Grand Rapids, Michigan
  - Colon and Rectal Surgery Associates Ltd, Saint Paul, Minnesota
  - Washington University School of Medicine - Barnes Jewish West, St Louis, Missouri
  - Colon & Rectal Surgery Inc, Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - Mt Sinai Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Methodist Hospital, Houston, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Fleshman JW, Beck DE, Hyman N, Wexner SD, Bauer J, George V; PRISM Study Group. A prospective, multicenter, randomized, controlled study of non-cross-linked porcine acellular dermal matrix fascial sublay for parastomal reinforcement in patients undergoing surgery for permanent abdominal wall ostomies. Dis Colon Rectum. 2014 May;57(5):623-31. doi: 10.1097/DCR.0000000000000106. PMID 24819103
- [Derived] Itani KM, Rosen M, Vargo D, Awad SS, Denoto G 3rd, Butler CE; RICH Study Group. Prospective study of single-stage repair of contaminated hernias using a biologic porcine tissue matrix: the RICH Study. Surgery. 2012 Sep;152(3):498-505. doi: 10.1016/j.surg.2012.04.008. Epub 2012 Jul 3. PMID 22763262

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 subjects failed eligibility to continue to protocol-specific surgery after randomization.
Groups:
- Strattice Fascial Inlay: Strattice placed as a fascial inlay to support the ostomy site
- Standard Ostomy Construction: Ostomy created in the standard fashion
Period: Overall Study
Arm/Group | Strattice Fascial Inlay | Standard Ostomy Construction
Started | 60 | 60
Completed | 40 | 35
Not Completed | 20 | 25

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis population is the 113 subjects in the Intent To Treat population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Strattice Fascial Inlay | Standard Ostomy Construction | Total
Number analyzed (Participants) | 55 | 58 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.25 (13.65) | 59.14 (14.36) | 59.7 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 30 | 29 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 48 | 57 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 55 | 58 | 113

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Parastomal Hernia in Subjects Undergoing Permanent Abdominal Wall Ostomy Creation With and Without Strattice Fascial Inlay.
Time Frame: 24 months
Population: Efficacy Evaluable Population (received assigned treatment, completed all protocol-required evaluations, no major protocol violations).
Measure: Number; unit: participants
Arm/Group | Strattice Fascial Inlay | Standard Ostomy Construction
Number analyzed (Participants) | 49 | 53
participants | 6 | 7

2. Secondary Outcome: Stoma Complications
Time Frame: 30 days
Reporting Status: Not Posted

3. Secondary Outcome: Stoma Complications
Time Frame: more than 1 month postoperatively
Reporting Status: Not Posted

4. Secondary Outcome: Stoma Quality of Life
Time Frame: Serially over 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Strattice Fascial Inlay | Standard Ostomy Construction
Serious Adverse Events (participants affected / at risk) | 37/55 | 37/58
Other Adverse Events (participants affected / at risk) | 54/55 | 55/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Strattice Fascial Inlay (N=55) | Standard Ostomy Construction (N=58)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Application Site Bleeding (General disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Acute Renal Failure (Renal and urinary disorders) | 3 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Malignant Tumour Excision (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Radiotherapy (Surgical and medical procedures) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Vesical Fistula (Renal and urinary disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Self Injurious Behaviour (Psychiatric disorders) | 0 | 1
Anal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Rectal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Crohn's Disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 | 0
Ileorectal Fistula (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 4 | 2
Ischiorectal Hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Proctitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 8
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Acinetobacter Bacteraemia (Infections and infestations) | 1 | 0
Administration Site Infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 2 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Pelvic Abscess (Infections and infestations) | 2 | 1
Perianal Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Urinary Tract Infection (Infections and infestations) | 3 | 0
Urosepsis (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 2 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complications (Injury, poisoning and procedural complications) | 7 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 3 | 6
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Open Wound (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Strattice Fascial Inlay (N=55) | Standard Ostomy Construction (N=58)
Anaemia (Blood and lymphatic system disorders) | 18 | 10
Tachycardia (Cardiac disorders) | 7 | 9
Abdominal Distension (Gastrointestinal disorders) | 13 | 9
Asthenia (General disorders) | 4 | 5
Abdominal Abscess (Infections and infestations) | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Abdominal Pain (Gastrointestinal disorders) | 20 | 22
Constipation (Gastrointestinal disorders) | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 2 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 3
Ileus (Gastrointestinal disorders) | 6 | 4
Intestinal Obstruction (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 29 | 30
Proctalgia (Gastrointestinal disorders) | 5 | 5
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 | 7
Vomiting (Gastrointestinal disorders) | 21 | 20
Chest Pain (General disorders) | 3 | 3
Fatigue (General disorders) | 9 | 15
Oedema Peripheral (General disorders) | 3 | 3
Pyrexia (General disorders) | 13 | 10
Cellulitis (Infections and infestations) | 3 | 4
Pneumonia (Infections and infestations) | 4 | 3
Postoperative Wound Infection (Infections and infestations) | 3 | 4
Sepsis (Infections and infestations) | 1 | 3
Urinary Tract Infection (Infections and infestations) | 13 | 13
Urosepsis (Infections and infestations) | 3 | 0
Wound Infection (Infections and infestations) | 3 | 2
Gastrointestinal Stoma Complications (Injury, poisoning and procedural complications) | 18 | 21
Incision Site Pain (Injury, poisoning and procedural complications) | 5 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 8 | 7
Procedural Pain (Injury, poisoning and procedural complications) | 3 | 5
Procedural Site Reaction (Injury, poisoning and procedural complications) | 13 | 12
Abnormal Breathing (Investigations) | 0 | 3
Oxygen Saturation Decreased (Investigations) | 1 | 5
Urine Output Decreased (Investigations) | 5 | 3
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 8 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Malnutrition (Metabolism and nutrition disorders) | 1 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Nervous system disorders) | 5 | 7
Headache (Nervous system disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 2 | 3
Confused State (Psychiatric disorders) | 1 | 5
Depression (Psychiatric disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 4 | 4
Haematuria (Renal and urinary disorders) | 2 | 6
Acute Renal Failure (Renal and urinary disorders) | 4 | 4
Urinary Incontinence (Renal and urinary disorders) | 1 | 3
Urinary Retention (Renal and urinary disorders) | 3 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Incisional Drainage (Surgical and medical procedures) | 4 | 2
Hypertension (Vascular disorders) | 4 | 2
Hypotension (Vascular disorders) | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less